CLINICAL TRIAL: NCT07080164
Title: Evaluation of Oral Health-Related Quality of Life In Patients With Conventional Complete Dentures Versus Mini-Implant Retained Overdentures: A Randomized Clinical Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yasmien Emad Eldeen, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1-1-2
Record Dates: First submitted 2025-07-15; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Complete Edentulism
Keywords: mini-implant overdentures ,OHRQoL ,RCT, Minimally invasive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- conventional dentures (Active Comparator)
  Interventions: Other: mini implant retained overdenture
- mini implant retained overdenture (Experimental): mini implant retained overdenture
  Interventions: Other: mini implant retained overdenture

INTERVENTIONS:
Other: mini implant retained overdenture — mini implant retained overdenture

SUMMARY:
Mini-implants have emerged as a practical and less invasive solution for the rehabilitation of edentulous mandibles, offering reduced surgical complexity, lower cost, and faster healing compared to conventional implants. These advantages make them especially suitable for elderly patients or those with systemic health concerns or limited bone volume. Despite their growing clinical use, evidence from well-designed randomized controlled trials evaluating the impact of mini-implant-retained overdentures on patients' oral health-related quality of life (OHRQoL) is still scarce. Establishing this evidence is crucial for guiding treatment decisions in resource-constrained settings and improving the standard of care for edentulous individuals. This research aims to provide high-quality data on the effectiveness of mini-implants in improving OHRQoL, as measured by OHIP-14, compared to conventional dentures./

ELIGIBILITY:
Inclusion Criteria:

* Completely edentulous mandible for a minimum period of 6 months Adult patients capable of understanding, cooperating, and providing informed consent Sufficient bone volume and interarch space in the anterior mandible to accommodate two mini-implants and overdenture attachments Good general health permitting minor oral surgical procedures Willingness to undergo follow-up visits and comply with study protocols

Exclusion Criteria:

* Systemic medical conditions that preclude implant surgery, including poorly controlled chronic diseases such as diabetes mellitus or disorders affecting bone metabolism.

Patients taking medications known to affect bone metabolism (e.g., bisphosphonates, corticosteroids) Patients with physical or mental disabilities that impair oral hygiene maintenance or compliance Heavy smokers (>10 cigarettes/day) Individuals unable or unwilling to attend scheduled follow-up or participate throughout the study duration Patients who can receive standard implants with no anatomical limitations

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
OHRQoL | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Oral and Dental Medicine Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided